CLINICAL TRIAL: NCT02496377
Title: Comparison of Preoperative Haemoglobin Level After Administration of Epoetin Alfa Associated With an Oral Versus Intravenous Iron Supplementation
Brief Title: Cross Iron (Comparative Randomized Oral Versus Systemic IRON)
Acronym: Cross Iron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9408; 2014-A00642-45 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-06-19; First posted 2015-07-14 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Allogenic Transfusion; Perioperative Anaemia; Knee Arthroplasty; Hip Arthroplasty
Keywords: Anaemia; Iron deficiency; Ferric carboxymaltose; Patient blood management; Hip arthroplasty; Knee arthroplasty
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — Epoetin Alfa; ferric carboxymaltose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Per Os Tardyferon (Active Comparator): EPO associated with Iron per os tardyferon before surgery. The oral group received 160 mg ferrous glycine sulfate daily during the month prior surgery, associated with 3 epoetin alpha (EPO) injections (40 000 IU subcutaneous on day - 21, day - 14 and day-7).
  Interventions: Drug: ferrous glycine sulfate Tardyferon; Drug: Epoetin Alfa
- Group 2: IV Ferinject (Experimental): EPO associated with Iron per IV Ferinject before surgery. The IV group received ferric carboxymaltose 1000 mg IV in 15 minutes one month before surgery, associated with 3 EPO injections.
  Interventions: Drug: Epoetin Alfa; Drug: ferric carboxymaltose Ferinject

INTERVENTIONS:
Drug: ferrous glycine sulfate Tardyferon
  Arms: Group 1: Per Os Tardyferon
Drug: Epoetin Alfa
Drug: ferric carboxymaltose Ferinject
  Arms: Group 2: IV Ferinject

SUMMARY:
Patients were recruited at the scheduled preoperative visit for hip or knee arthroplasty. If the haemoglobin (Hb) level was below 13 g/dl with no contraindication to iron supplementation the patients were randomized to the oral or intravenous (IV) group. The oral group received 160 mg ferrous glycine sulfate daily during the month prior surgery, associated with 3 epoetin alpha (EPO) injections (40 000 IU subcutaneous on day - 21, day - 14 and day-7). The IV group received ferric carboxymaltose 1000 mg IV in 15 minutes one month before surgery, associated with 3 EPO injections. Primary efficacy endpoint was the change in Hb level from the day of the preoperative visit to the day before surgery (day-1). Secondary endpoints comprised the Hb level on day 3 and 5 after surgery, allogenic transfusion during and after surgery, and the change in iron indices from the day of the preoperative visit to day - 1.

ELIGIBILITY:
Inclusion criteria:

* unilateral prothetic orthopaedic surgery scheduled
* age > 18
* weight > 50 kg
* hemoglobin rate: 10 g/dl ≤ Hb <13 g/dl

Exclusion criteria:

* bilateral arthroplasty
* EPO contraindication
* generalized infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08-29 (Actual); Primary Completion 2016-10-16 (Actual); Study Completion 2016-10-16 (Actual)

PRIMARY OUTCOMES:
Compare Hb level after treatment with EPO associated with iron treatment by oral or intravenous route | the day before surgery (day - 1)

SECONDARY OUTCOMES:
Hb level | before iron treatment, then the day before surgery (day - 1) based on reference iron balance
number of red blood cells | during surgery and 3 days after surgery
the change in iron indices | before iron treatment and after iron treatment the day before surgery (day - 1)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BIBOULET, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Hôpital Lapeyronie - Département Anesthésie Réanimation A, Montpellier, France